CLINICAL TRIAL: NCT04990258
Title: A 24-month Real Life PErsistence Efficacy and Safety Study in IBD Patients in REMission Switched From Intravenous Infliximab to Subcutaneous Infliximab CT-P13 Remsima®SC
Acronym: PEREM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Celltrion (Industry)
Responsible Party: Sponsor
Other Study IDs: GT-2021-02
Record Dates: First submitted 2021-06-14; First posted 2021-08-04 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD UC
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Subcutaneous infliximab CT-P13 Remsima®SC — Patients will be switched from IV infliximab into subcutaneous infliximab Remsima®SC 120 mg.

SUMMARY:
Descriptive: A 24-month multicentre, observational, prospective cohort study. Population: IBD Patients under stable clinical and biological remission Study treatments: Patients who will be proposed to switch, or who have just switched, from the intravenous originator Remicade® or one of its biosimilars to the subcutaneous infliximab Remsima®SC as part of routine care. All consecutive patients in IBD centers participating in the study will be proposed to participate in the study during their regular outpatients' visits.

Objectives:The primary objective of PEREM study is to determine the rate of persistence of subcutaneous infliximab at 48 weeks after switching from IV infliximab to subcutaneous infliximab Remsima®SC.

DETAILED DESCRIPTION:
Number of patients: 400 patients in approximatively 40 sites in France Recrutment period: The trial duration for each patient will be 2 years Main Endpoint:The primary endpoint is to assess the rate of persistence of subcutaneous infliximab at month 12 after switching from IV infliximab to SC infliximab Remsima®SC.

Secondary Endpoint:

* Percentage of patients on steroid free clinical remission at week 96 after switch. Steroid-free Clinical Remission (CR) is defined as a Harvey Bradshaw Index (HBI) score≤4 CD patients and a Partial Mayo Score (PMS) ≤2 with each sub-score of 1 or less for UC. When HBI scoring will be infeasible (stoma, pouch), evaluation of clinical remission will be estimated by stoma emptying count and/or by the physician global assessment (Sturm 2019) Patients having discontinued subcutaneous infliximab Remsima®SC therapy whatever the reason during the 24 months of follow-up as well as patients referred to disease-related surgery and patients lost to follow-up before month 24 will be considered as failure to subcutaneous infliximab Remsima®SC therapy (intention to treat analysis) and will be classified in the group of patients having failed to maintain steroid free clinical remission under infliximab Remsima®SC during the whole study period.
* Percentage of patient Reported Outcomes PRO2 rates at inclusion, months 3, 6, 12 and 24
* Percentage of biological remission rates (FC <250 μg/g, CRP <5 mg/L) at inclusion, month 3, 6, 12 and 24.
* Percentage of clinical relapse free rates at inclusion, month 3, 6, 12 and 24
* Percentage of loss of response rates at inclusion, month 3, 6, 12 and 24
* Percentage of clinical response and remission at inclusion, month 3, 6, 12 and 24
* Mean change from baseline in HBI or PMS, and mean change from baseline in CRP and fecal calprotectin
* Proportion of patients with positive antibodies (IFX, ANA) comparing therapy with intravenous or one of its biosimilars original and subcutaneous infliximab Remsima®SC
* Measure adherence to subcutaneous infliximab Remsima® switch based on pharmacy data during the follow-up with Medication Possession Ratio (MPR ).
* Twelve-month cumulative surgery rates
* Hospitalization rate at month 24
* Cumulative infection rate at month 24
* Cumulative SC reactions at month 24
* Discontinuation of subcutaneous infliximab therapy cumulative rates at month 24
* Incidence of specific anti-drug antibodies detected during the study

ELIGIBILITY:
Inclusion Criteria:

* • Male or female subjects who are more than 18 years of age, on the day of signing informed consent.

  * Patient affiliated to the health insurance system.
  * Documented diagnosis of CD or UC established based on standard clinical, endoscopic, and histological criteria.
  * CD or UC remission defined per clinical assessment as a Harvey Bradshaw Index (HBI) score ≤4 for CD patients and a Partial Mayo Score (PMS) ≤2 with each sub-score of 1 or less for UC and/or according to ECCO classification within previous 6 months.
  * Currently treated with IV infliximab: originator or biosimilars.
  * Patients agreeing to switch from IV to SC formulation or who have already switched since maximum 3 months.
  * Receiving or not the concomitant following drugs (but must remain on stable dose for 12 weeks):
* Oral 5-aminosalicylates (5ASA) compounds or rectal formulations of 5ASA provided the dose to be stable at least 4 weeks before switching.
* Azathioprine, 6-MP or methotrexate provided the dose has been stable for 4 weeks prior to inclusion (dose must remain stable for 10 weeks after switching).

  * Each patient is required to provide written informed consent to be included in the study.

Exclusion Criteria:

* Current use of vedolizumab or ustekinumab
* Current use of JAK inhibitors or S1P modulators
* Current use of steroids or within the last three months for IBD
* Treatment with any investigational agent in the past 30 days or five half-lives prior to the inclusion visit
* Current CD abscess
* Active clinically significant infection or HIV, Hep B, Hep C, untreated tuberculosis
* Female subjects with pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age ≥ 18 ans, CD patients (HBI ≤4) or UC patients (PMS ≤2) with established diagnosis > 6 months treated with Infliximab IV, agreeing to switch from IV to SC formulation or who have just switched to subcutaneous infliximab Remsima®SC as part of routine care
Sampling Method: Non-Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Subcutaneous infliximab dosage after switch | Month 12
  To describe subcutaneous infliximab persistence after the switch from IV infliximab originator Remicade® or one of its biosimilars to SC infliximab (Remsima®SC) at month 12.
Efficacy of Subcutaneous infliximab treatment in clinical remission | Month 24
  Steroid-free clinical remission 24 months after switching
Safety of subcutaneous infliximab treatment | Month 24
  Proportion of participants with treatment-related adverse events for a period of 24 months after switching

SECONDARY OUTCOMES:
Ratio efficacy of SC Infliximab in clinical remission | Month 24
  Percentage of patients on steroid free clinical remission at month 24 after switch.
  * Steroid-free Clinical Remission (CR) is defined as a Harvey Bradshaw Index (HBI) score≤4 for CD patients and a Partial Mayo Score (PMS) ≤2 with each sub-score of 1 or less for UC.
  * When HBI scoring will not be feasible (stoma, pouch), evaluation of clinical remission will be estimated by physician global assessment.
  * Patients having discontinued subcutaneous infliximab therapy whatever the reason during the 12 months of follow-up as well as patients referred to disease-related surgery and patients lost to follow-up before month 24 will be considered as failure to subcutaneous infliximab Remsima®SC therapy (intention to treat analysis) and will be classified in the group of patients having failed to maintain steroid free clinical remission under subcutaneous infliximab Remsima®SC during the whole study period
Loss of response to infliximab SC treatment | Month 12
  Percentage of patients who switch back to originator previous therapy IV infliximab at month 12 after switching from IV infliximab to SC infliximab Remsima®SC in IBD patient
Efficacy of SC Infliximab treatment on patient quality of life | Month 12
  Percentage of PRO2 response and remission at month 12
Efficacy of SC Infliximab treatment in biological remission | Month 12
  Percentage of biological remission rates (FC <250 μg/g, CRP <5 mg/L) at month 12
Efficacy of SC Infliximab treatment in preventing relapse | Month 12
  Percentage of clinical relapse free rates at month 12.
Efficacy of SC Infliximab treatment in preventing loss of respone | Month 12
  Percentage of loss of response rates at month 12
Loss of clinical response | Month 3
  Percentage of clinical response and remission at month 3
Disease activity | Month 24
  Mean change from baseline in
  * For Crohn Disease: HBI( Harvey Bradshaw Index):
  * For Ulcerative Colitis: PMS ( Partial mayo score)
  * Biological criteria
    * CRP (mg/l): Remission < 5 mg CRP in 1 litre of blood and
    * fecal calprotectin ( μg/g ) : Remission < 250 μg of fecal calprotectin in 1 g of stool
  HBI score, PMS score, CRP and Calprotectin feacal will be combined to report the disease activity (this outcome is is expressed without units)
Treatment adherence | Month 24
  Proportion of patients with positive antibodies (IFX, ADA) comparing therapy with original and SC infliximab.
Medication Possession Ratio (MPR) | Month 24
  Adherence to biosimilar switch during the follow-up: MPR ratios.

CONTACTS AND LOCATIONS:
Locations (1):
- Nicolas Mathieu, Grenoble, France